CLINICAL TRIAL: NCT02784730
Title: A Randomized, Multicentre, Comparative Phase III Study of Catheter-related Complications of an Iterative PICC Placement vs a Long-term PAC in Patients With Breast Cancer
Brief Title: Iterative PICC Placement Versus Long Term Device
Acronym: PICC One Day
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Changes of the standard adjuvant treatment which does not allow an iterative PICC placement
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government); C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PICC One Day 01 (ET15-123); 2015-A01822-47 (Other: ID-RCB number)
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; peripherally inserted central catheter; implantable device; randomized controlled trial; iterative placement; Catheterization, Central Venous
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iterative PICC placement (Experimental): New PICC placement at each chemotherapy cycle (removed after treatment administration)
  Interventions: Procedure: Iterative PICC placement
- Long term implantable device (Active Comparator): Port-a-cath inserted prio first chemotherapy cycle and maintained throughout the study
  Interventions: Procedure: Long term PAC placement

INTERVENTIONS:
Procedure: Iterative PICC placement — Intervention is the catheterisation strategy (not the device)
  Arms: Iterative PICC placement
Procedure: Long term PAC placement — Intervention is the catheterisation strategy (not the device)
  Arms: Long term implantable device

SUMMARY:
Peripherally Inserted Central Catheter (PICC) and port-a-cath (PAC) are the most commonly medical devices used for the administration of chemotherapy.

Placement of these devices via central venous access is sometimes responsible for complications.

The incidence of these complications is correlated with the device holding time.

A strategy of iterative PICC placement could significantly reduce these complications.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years old;
* Breast cancer diagnosis histologically proven , for any histological subtypes;
* 4 or 6 indication of neoadjuvant or adjuvant chemotherapy; according to hormonal status and HER2 of the tumors, the patient may be treated concomitantly with hormone therapy and / or trastuzumab; Nota Bene: treatment protocol adopted will imperatively be administered in 3-week cycles.
* Central venous access indication;
* Ability to understand and willingness to comply with the study monitoring;
* Affiliated to the French social security system;
* Informed Consent dated and signed, indicating that the patient has been informed of all pertinent aspects of the study before inclusion.

Exclusion Criteria:

* Any contraindication for placement of a central venous catheter ( hemostasis disorders , active infection treated with antibiotics , ...);
* Patient who can't stop anti -vitamin K treatment ( AVK ) ( a relay by Heparin Low Molecular Weight (LMWH) is possible);
* History of central access, regardless of the indication;
* Any active disease other than cancer pathology , requiring repeated administration of intravenous therapy ;
* Patient deprived of liberty;
* Not monitoring for social, geographical, psychological or family reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Compare complication rate for iterative placement (PICC) versus long term placement (PAC). | 6 months after randomization
  Complication rate will be defined by the proportion of patients with at least one of the following complications from the date of randomization to the end of the study:
  pneumothorax , hemothorax ,veinous thrombosis, migration or expulsion of the device, fissure or rupture of the catheter, catheter obstruction, extravasation.

SECONDARY OUTCOMES:
Success rate for each strategy | 6 months after randomization
  Success rate will be determined with the proportion of patients in whom the allocation strategy was conducted until the end of the last cycle of chemotherapy
Description of failure causes for each strategy | 6 months after randomization
  Causes of failures will be described
Level of pain for each strategy | At Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1
  Level of pain will be assessed with the verbal scale rated from 0 to 10
Quality of Life in both arms | At Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1
  Quality of Life will be assessed with the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hervé ROSAY, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Julien GAUTIER, Lyon, France

IPD SHARING:
Plan to Share IPD: No